CLINICAL TRIAL: NCT03899233
Title: Comparing Tranexamic Acid Microinjection Alone Versus Its Combination With Fractional Carbon Dioxide Laser in Melasma Treatment
Brief Title: Tranexamic Acid vs. Combination With Fractional Carbon Dioxide Laser in Melasma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Raafat Said, Lecturer of Dermatology Department, Faculty of Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Melasma treatment
Record Dates: First submitted 2019-03-21; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Melasma
Keywords: Melasma; Tranexamic acid; Fractional CO2 laser
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: Each participate will be assigned to both arms (split face manner). One half of the face will be assigned to Tranexamic acid alone and the other side of the face will be assigned to combined Tranexamic acid and Fractional CO2 laser. Both sides of the face will take the same time of treatment and will be assessed at the same time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional CO2 laser combined with Tranexamic acid (Active Comparator): one side of the face of all participants will be subjected to low power fractional CO2 laser with a power of 12 watts, spacing 800 micrometer (7.3% density), and dwell time 300 microsecond for 3 sessions every 6 weeks. In addition to Tranexamic acid intradermal microinjections using tranexamic acid 500mg/5ml ampoules, the dose of 1ml syringe with 100mg/ml with maximum of 4ml per session, on the 2nd and the 4th week of each laser session. With total treatment time for each patient of 4 months and another month free of sessions for followup.
  Interventions: Device: Fractional CO2 laser; Drug: Tranexamic acid intradermal microinjections
- Tranexamic acid alone (Active Comparator): the other side of the face of all participants will be subjected Tranexamic acid intradermal microinjections using tranexamic acid 500mg/5ml ampoules, the dose of 1ml syringe with 100mg/ml with maximum of 4ml per session, every 2 weeks for 4 months then another month free of sessions for followup.
  Interventions: Drug: Tranexamic acid intradermal microinjections

INTERVENTIONS:
Device: Fractional CO2 laser — Low power fractional CO2 laser with a power of 12 watts, spacing 800 micrometer (7.3% density), and dwell time 300 microsecond
  Arms: Fractional CO2 laser combined with Tranexamic acid
Drug: Tranexamic acid intradermal microinjections — Tranexamic acid 500mg/5ml ampules

SUMMARY:
The objective of this study is to assess and compare the efficacy of tranexamic acid intradermal microinjection alone versus its combination with low power fractional CO2 laser in a sequential pattern.

In all participants one half of the face will be randomly assigned to low power fractional CO2 laser while other side to Tranexamic acid intradermal microinjections on the 1st session. This split face session will be repeated every six weeks for 3 sessions.

In addition, Tranexamic acid intradermal microinjections will be applied for full face at the 2nd and 4th week of each split face session.

The response will be evaluated by the Melanin and erythema Indices which will be measured using reflectance spectrophotometer, Dermoscopy and photography before starting the study, two and four weeks after the last session. The sessions will take 4 months for each patient and another one month free of sessions for follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral symmetrical facial melasma

Exclusion Criteria:

* Pregnancy and lactation.
* Patients taking oral contraceptive pills or hormonal replacement therapy at the time of the study or during the past 12 months.
* Concomitant use of anticoagulants.
* Bleeding disorders.
* Personal or family history of deep venous thrombosis or thromboembolic events.
* Scarring and keloid tendency.
* Active skin infection, active Herpes simplex virus.
* History of Post-inflammatory hyperpigmentation.
* History of photosensitivity or photosensitizing medication as sulfonamides tetracycline,retinoids, bleaching creams, peeling and laser two months before the study.
* Occupational sun exposure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Melanin and Erythema indices change from baseline | baseline, 18 weeks and 20 weeks
  Comparing the effect of Tranexamic acid intradermal microinjection alone versus its combination with low power fractional CO2 laser in a sequential pattern on melasma improvement by measuring the Melanin and erythema Indices (MI and EI) using reflectance spectrophotometer before starting the study, two and four weeks after the last session.
Dermoscopic features change from baseline | baseline, 18 weeks and 20 weeks
  Comparing the effect of Tranexamic acid intradermal microinjection alone versus its combination with low power fractional CO2 laser in a sequential pattern on melasma improvement by Dermoscopy before starting the study, two and four weeks after the last session.

REFERENCES:
- [Background] Tawfic SO, Abdel Halim DM, Albarbary A, Abdelhady M. Assessment of combined fractional CO2 and tranexamic acid in melasma treatment. Lasers Surg Med. 2019 Jan;51(1):27-33. doi: 10.1002/lsm.23032. Epub 2018 Nov 15. PMID 30431171
- [Background] Trelles MA, Velez M, Gold MH. The treatment of melasma with topical creams alone, CO2 fractional ablative resurfacing alone, or a combination of the two: a comparative study. J Drugs Dermatol. 2010 Apr;9(4):315-22. PMID 20514787
- [Background] Jalaly NY, Valizadeh N, Barikbin B, Yousefi M. Low-power fractional CO(2) laser versus low-fluence Q-switch 1,064 nm Nd:YAG laser for treatment of melasma: a randomized, controlled, split-face study. Am J Clin Dermatol. 2014 Aug;15(4):357-63. doi: 10.1007/s40257-014-0080-x. PMID 24858737
- [Background] Saki N, Darayesh M, Heiran A. Comparing the efficacy of topical hydroquinone 2% versus intradermal tranexamic acid microinjections in treating melasma: a split-face controlled trial. J Dermatolog Treat. 2018 Jun;29(4):405-410. doi: 10.1080/09546634.2017.1392476. Epub 2017 Nov 9. PMID 29027510